CLINICAL TRIAL: NCT01353768
Title: Medical Record Review and Data Abstraction for Pediatric, Adolescent and Pregnant Patients Treated With IV Zanamivir in the Relenza Compassionate Use Program
Brief Title: Zanamivir Aqueous Solution Compassionate Use Program Retrospective Chart Review Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115008
Record Dates: First submitted 2011-04-21; First posted 2011-05-16 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Respiratory Tract
Keywords: Influenza
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: zanamivir aqueous solution administered previously as part of the Compassionate Use Program
  Interventions: Other: retrospective chart review

INTERVENTIONS:
Other: retrospective chart review — retrospective chart review

SUMMARY:
GSK is conducting a global retrospective chart review of patients treated with zanamivir as part of the Compassionate Use Program (CUP), in an effort to collect as much information as possible on the use of this investigational drug. The retrospective chart review is intended to gain a better understanding of the safety profile of investigational zanamivir and of clinical outcomes in the large number of patients treated outside of a clinical trial setting.

DETAILED DESCRIPTION:
This is an observational, retrospective, multi-centre, cohort data collection study.

The CUP retrospective review study has been designed to collect safety and clinical outcome data from pediatric and pregnant patients (collectively referred to as the "Tier 1" cohort) treated globally within the CUP during the 2009/2010 pandemic (from May 2009) through 31 January 2011. The study will also attempt to collect data from other adult patients (referred to as the "Tier 2" cohort) who were treated at sites identified as having Tier 1 patients.

The treating physician at each site will receive a letter from the GSK medical director inviting him/her to participate in the retrospective chart review study. Physicians (or their delegates) who agree to participate will receive study-related documentation [including the protocol and case report form (CRF)] to orient the site to the study details and CRF. For the purposes of this study, the term "site" generally refers to a hospital where in-patient treatment was provided.

The retrospective chart review will be monitored via remote visits by telephone. The interviewer will be a Kendle associate assigned to the study who will not have direct access to the patient's source documents or medical records during conduct of the study. The physician/delegate will review the patient's chart and record data on a paper CRF. The CRF will be in the English language. Site personnel will mail completed CRFs to Kendle. Kendle will review the CRF for data quality, and conduct a remote monitoring visit via telephone to address any data queries, if required. No visits to participating sites are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric or pregnant patients that received zanamivir aqueous solution as part of the Compassionate Use Program from May 2009 through 31 January 2011 (Tier 1 cohort).
2. Adult patients (Tier 2 cohort) that received zanamivir aqueous solution as part of the Compassionate Use Program from May 2009 through 31 January 2011, treated at the same site as a Tier 1 patient.

Exclusion Criteria:

1. Adult patients that received zanamivir aqueous solution at non-Tier 1 sites.
2. Pediatric or pregnant patients that received zanamivir aqueous solution as part of the Compassionate Use Program after 31 January 2011.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 350 patients previously treated with zanamivir aqueous solution as part of the CUP, at an estimated 100 sites in over 15 countries are targeted for participation. Medical information on safety and clinical outcomes from Tier 1 and Tier 2 patients will be collected within this retrospective chart review study.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mortality | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients who died

SECONDARY OUTCOMES:
Other anti-influenza therapies | for duration of influenza-related hospitalization, an expected average of 5 weeks
  Number of patients who received other anti-influenza therapies
Chest X-ray abnormalities | within 1-2 days of hospital admission or symptom onset
  Number of patients with abnormal findings
Resistance to zanamivir | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients with documentation of resistance
Other infections | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients with diagnosis of other infections
Complications of influenza | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients with complications of influenza
Ventilation/Oxygenation | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients requiring ventilation support or supplemental oxygen
Concomitant Medications | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients receiving antibiotic/, antifungal/, orticosteroids, or inotropic medications
Treatment emergent events | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients experiencing a treatment emergent event
Hemodialysis/Renal Replacement Therapy | for duration of influenza-related hospitalization, an expected average duration of 5 weeks
  Number of patients receiving hemodialysis or renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register